CLINICAL TRIAL: NCT04346745
Title: Developing a Culturally-sensitive Volunteering Program to Reduce Stress of Dementia Caregivers in Chinese American Communities
Brief Title: Volunteering Program for Chinese Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS3969
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Caregiver Burnout
Keywords: Chinese; Volunteering; Peer mentoring; dementia caregivers; mental health; stress
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group will receive intervention of a peer mentoring program plus usual services they could receive from community agencies.
  Interventions: Behavioral: Peer Mentoring Program
- Control group (No Intervention): The control group received a package of educational materials on knowledge of dementia, caregiving skills.

INTERVENTIONS:
Behavioral: Peer Mentoring Program — The Peer Mentoring Program (PMP) is a 3-month intervention to provide one-on-one mentoring support via phone calls to reduce the stress of Chinese dementia caregivers. The PMP will address the following topics: cultural beliefs about dementia and family caregiving, culturally effective coping strategies, and culturally appropriate social support.
  Arms: Treatment group

SUMMARY:
Although many older Chinese Americans are expected to need intensive care because of cognitive impairment, a large gap exists in development of culturally sensitive interventions to reduce stress among caregivers in Chinese American communities. This research project will develop and pilot test a culturally sensitive intervention, the peer mentoring program (PMP), which is informed by the sociocultural stress and coping model. This project will generate preliminary data for a larger randomized controlled trial for efficacy or effectiveness testing of PMP, which is an innovative intervention to support dementia among Chinese Americans, by empowering the existing human resources of experiential caregivers in the same ethnic community.

DETAILED DESCRIPTION:
Providing care for a family member with Alzheimer's disease and related dementia (ADRD) negatively affects caregivers' physical and mental health.Despite numerous studies on developing interventions for ADRD family caregivers of Caucasian Americans, it is not clear what interventions are effective in reducing the stress of family caregivers of Asian Americans. The purpose of this study is to develop a culturally sensitive and effective intervention to reduce the stress of dementia caregivers of Chinese Americans. It is necessary to prioritize Chinese American ADRD caregiving research because of: (a) the increasing needs of ADRD caregivers of Chinese Americans, the largest and fastest-growing ethnic group of Asians in the United States; (b) erroneous conclusions about Chinese American health in current research and policy practices due to omission, aggregation, and extrapolation; (c) health inequality issues ignored by the "model minority" stereotype of Asian Americans in general; (d) mental health vulnerabilities of older Chinese Americans; and (e) unresolved challenges of Chinese American caregivers such as lack of health literacy, concerns about stigma, failure to maintain family harmony, social isolation, and barriers to accessing culturally competent services. Given these concerns and the lack of health professionals who can speak Chinese and understand Chinese culture and norms, this study aims to develop a peer mentoring program to support dementia caregivers by empowering the human resources of experiential caregivers in Chinese American communities.

Informed by the sociocultural stress and coping model and relevant empirical evidence, the investigators designed the Peer Mentoring Program (PMP) to train and monitor experiential caregivers in providing mentoring support for caregivers in the same ethnic community. Experiential caregivers in the same ethnic community could understand the caregiving journey embedded in Chinese cultural values and the international migration experience. In the PMP, experiential caregivers will be hired and trained as volunteer peer mentors and monitored in providing mentoring support to dementia caregivers to address cultural beliefs about dementia and family caregiving, develop culturally effective coping strategies, and enhance culturally appropriate social support. The intervention is promising given the needs of Chinese caregivers, positive results of a previous trial in a senior volunteer program in Chinese Americans communities, benefits of volunteering for older adults, preliminary analysis results of data from our pilot study (70% Chinese caregivers reported a desire to receive peer mentoring support), and the potential of developing a cost-effective and sustainable intervention that could be applied in other racial and ethnic minority communities.

This proposed study will use a community-based participatory research (CBPR) approach based on a partnership of multidisciplinary researchers, health professionals, family caregivers and older volunteers in NYC to accomplish Stage 0 (Aim1) and Stage I (Aims 2 and 3) for behavioral intervention development and to develop Stage II and/or Stage IV (Aim 3).

Aim 1: To study the challenges and enablers of successful caregiving for persons with ADRD in Chinese American communities in New York City (NYC). The investigators will analyze recently collected data from in-depth interviews and questionnaire-based surveys to identify robust challenges, barriers, resources, and successful coping strategies among these caregivers, which will help develop the PMP intervention manual.

Aim 2: To develop the PMP intervention protocol. Using the analysis results from Aim 1 in collaboration with multidisciplinary researchers and professionals, I will develop the volunteer training manual, intervention protocol, and screening and evaluation tools.

Aim 3: To examine the feasibility and acceptability of PMP. A pilot randomized clinical trial of five volunteers and 30 caregivers (15 to intervention, 15 to control) will be conducted. Qualitative and quantitative data from caregivers, volunteers, and professional collaborators will be collected to evaluate feasibility and acceptability of recruitment, randomization, intervention adherence, treatment fidelity, and administration of measures. Based on the results of feasibility and acceptability test, The investigators will refine the intervention and inform a subsequent larger randomized control trial (RCT) to initiate an efficacy or hybrid stage of intervention development.

ELIGIBILITY:
Inclusion Criteria:

The caregivers will be recruited if they:

* self-identify as Chinese
* are 21 years old or older
* speak Mandarin or Cantonese Chinese
* provide care to a family member with dementia or cognitive impairment related to dementia for 10 hours or more a week
* are interested in receiving peer mentoring
* report moderate to severe caregiver burden
* can access a telephone and communicate via phone call.

Inclusion Criteria:

The volunteer mentors will be recruited if they:

* are 50 years old or older
* self-identify as Chinese
* speak Mandarin or Cantonese Chinese
* have experience providing care to a family member with dementia or cognitive impairment related to dementia
* can access a telephone and communicate via phone call
* can attend volunteering training in person
* agree to volunteer as a mentor with minimal financial compensation
* agree to the time commitment required by the program.

Exclusion Criteria for both groups:

* do not self-identify as Chinese
* do not speak Mandarin or Cantonese Chinese

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Liu, PhD, Principal Investigator — Baylor University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Cheung ESL, Lou Y, Wu B. A peer mentoring program for Chinese American dementia caregivers: a pilot randomized controlled trial. Aging Ment Health. 2024 Nov;28(11):1479-1488. doi: 10.1080/13607863.2024.2346599. Epub 2024 May 2. PMID 38695396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 19 | 19
Completed | 18 | 16
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.11 (11.74) | 67.16 (13.57) | 67.13 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 19 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
loneliness [Mean (Standard Deviation); unit: units on a scale] | 4.74 (2.31) | 4.18 (1.5) | 4.46 (1.94)
caregiver burden [Mean (Standard Deviation); unit: units on a scale] | 22.63 (9.96) | 23.26 (6.64) | 22.95 (8.36)
caregiving competency [Mean (Standard Deviation); unit: units on a scale] | 13.08 (1.93) | 13.00 (1.91) | 13.04 (1.90)
Depressive symptoms [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms were measured by the 10-item Center for Epidemiological Studies Depression Scale (Andresen et al., 1994). Caregivers reported their depressive symptoms in the past week on a 4-point scale (from 0 = rarely or none of the time to 3 = most or all of the time). The summed scores ranged from 0 to 30, and higher scores indicated higher levels of depressive symptoms (Cronbach's α = .86).
  units on a scale | 10.63 (7.95) | 8.79 (6.45) | 9.71 (7.20)

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Burden Score at Month 3 and Month 9
Description: This outcome will be measured by Zarit's Burden Interview (ZBI). ZBI contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). In general, higher score indicates higher levels of burden. The full summed score ranges from 0 to 88, with higher scores indicating higher levels of burden (Cronbach's α = .80).
Time Frame: Month 3, Month 9
Population: Four participants (1 in treatment group and 3 in control group) withdrew from the study before data was collected at Month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 16
units on a scale
  Month 3 | 23.73 (10.38) | 25.56 (7.80)
  Month 9 | 21.41 (11.89) | 27.67 (8.00)

2. Primary Outcome: Caregiver's Depression at Month 3 and Month 9
Description: Depressive symptoms were measured by the 10-item Center for Epidemiological Studies Depression Scale (Andresen et al., 1994). Caregivers reported their depressive symptoms in the past week on a 4-point scale (from 0 = rarely or none of the time to 3 = most or all of the time). The summed scores ranged from 0 to 30, and higher scores indicated higher levels of depressive symptoms (Cronbach's α = .86).
Time Frame: Month 3, Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 16
units on a scale
  Month 3 | 12.48 (7.56) | 13.00 (7.69)
  Month 9 | 9.61 (7.78) | 11.88 (6.62)

3. Primary Outcome: Caregiving Competency at Month 3 and Month 9
Description: Caregiving competency was measured by the Caregiving Competence Scale. It is a 4-point Likert (not at all, just a little, somewhat, very much) scale including four questions: How do you believe that you've learned to deal with very difficult situations? How much do you feel that all in all, you're a good caregiver? How competent do you feel? How self-confident do you feel? We summed the scores of four items with higher scores indicating larger competence (Cronbach's alpha=0.62). The range of the score is 0-16.
Time Frame: Month 3, Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 16
units on a scale
  Month 3 | 12.44 (2.41) | 13.00 (1.86)
  Month 9 | 13.00 (3.61) | 12.5 (2.85)

4. Primary Outcome: Loneliness at Month 3 and Month 9
Description: Loneliness was assessed by the Revised-University of California at Los Angeles Loneliness Scale. Caregivers rated their feelings of lacking companionship, left out of life, and isolation from others respectively on a 3-point scale (hardly ever, sometimes, often). We added up scores for the three questions to produce a continuous variable ranging from 0 to 6, with higher scores indicating higher levels of loneliness (Cronbach's alpha = 0.80).
Time Frame: Month 3, Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 16
units on a scale
  Month 3 | 4.56 (2.04) | 5.44 (2.00)
  Month 9 | 5.11 (2.32) | 5.31 (2.47)

ADVERSE EVENTS:
Time Frame: 9 months
Description: This is a behavioral intervention study. There is minimal risk of adverse events.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT04346745/Prot_SAP_000.pdf